CLINICAL TRIAL: NCT04086589
Title: Exploratory Pilot Study to Discover Genes That Restore the Molecular Circadian Rhythm
Brief Title: Restoring Molecular Circadian Rhythm
Status: Suspended | Type: Observational
Why Stopped: COVID-19
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 832866
Record Dates: First submitted 2019-08-19; First posted 2019-09-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Young; Healthy Elderly
Keywords: healthy, young, elderly
MeSH Terms: interventions — Observation; Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young: Observational study without intervention
  Interventions: Other: Observational study without intervention
- Elderly: Observational study without intervention
  Interventions: Other: Observational study without intervention

INTERVENTIONS:
Other: Observational study without intervention — Observational study without intervention

SUMMARY:
The goal is to address the mechanisms that account for alteration of circadian rhythms with age. As the blood of aged individuals can produce this alteration, the investigators propose to use such blood samples to "age" circadian rhythms in cultured cells. The investigators will verify aged blood-dependent alteration of rhythms and then conduct molecular screens to reverse this decline. If the investigators identify specific genes that can restore molecular circadian rhythm in vitro, the investigators will explore these in animal models (Drosophila, mouse).

ELIGIBILITY:
Inclusion Criteria:

* General good health with the following conditions permissible

  * cardiovascular risk prevention, intake of low dose aspirin,
  * hypertension, intake of beta-blockers, ACE inhibitors, diuretics, calcium channel blockers
  * hypercholesterinemia, intake of statins
* Cases: 70-85 years of age
* Controls: 20-35 years of age
* Patients must be able to read and understand English
* Participants must sign the informed consent form
* Participants must have a wrist-actigraphy-based average TST (total sleep time) ≥ 6 hours per night (measured over 7 consecutive days) occurring between 22:00 - 08:00

Exclusion Criteria:

* Known history of severe psychiatric or cognitive conditions, for example mania, schizophrenia, or mental retardation
* Shift work, defined as recurring work between 22:00-05:00
* History of clinically significant obstructive sleep apnea
* Transmeridian travel across ≥2 time zones in the two weeks prior to the blood draws and one week after,
* > 2 drinks of alcohol per day
* Use of illicit drugs

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparent healthy volunteers
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Delta of period length measured in hh:mm between in vitro cycling fibroblasts incubated with serum collected from cases (elderly adults) versus controls (young adults) | Time point 14:00 Hours
  To determine if serum collected from young versus old healthy study participants have a differential effect on the expression of circadian rhythms in an in vitro culture of a fibroblast cell line
Delta of phase measured in HH:mm between in vitro cycling fibroblasts incubated with serum collected from cases (elderly adults) versus controls (young adults) | Time point 14:00 Hours
  The primary endpoint will be the difference in phase angle in vitro between cycling fibroblasts and incubated with serum collected from cases (old adults) versus controls (young adults)

SECONDARY OUTCOMES:
Chronotype | 4 weeks
  Assessed per survey; chronotypes per Munich Chronotype questionnaire are extreme early type, moderate early type, slight early type, normal type, slight late type, moderate late type, extreme late type
Acrophase | 7 days
  Clock hour of peak physical activity averaged from 7 or more days of actigraphy
Physical activity | 7 days
  Vector magnitude of physical activity averaged from 7 or more days of actigraphy
Sleep quantity | 7 or more days
  Hours of sleep averaged from 7 or more days of actigraphy
Sleep quality: actigraphy | 7 days
  Sleep fragmentation averaged from 7 or more days of actigraphy
Ambient light exposure | 7 days
  Ambient light exposure averaged from 7 or more days of actigraphy
Heart rate variability | 24 hours
  Heart rate variability (RR intervals) averaged from 24 hours of BioPatch
Saliva cortisol | 24 hours
  Difference in concentrations of cortisol measured in saliva between morning versus evening

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skarke, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided